CLINICAL TRIAL: NCT03771079
Title: Evaluation of MassArray Platform Versus Illumina Miseq for the Detection of Driver Mutations in Hematological Malignancies
Brief Title: MS Detection of Somatic Mutations in Hematological Malignancies
Acronym: MAHM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7259
Record Dates: First submitted 2018-12-05; First posted 2018-12-10 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Hematological Malignancy
Keywords: Hematological Malignancy; mutations; NGS sequencing; mass spectrometry
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Detection of somatic mutations in hematological malignancies is now routinely assessed by NGS sequencing. This powerful approach is nevertheless time consuming and its costs represent limitation for its availability. An original approach is now available, using mass spectrometry (MS). In this study the analytical performance of both methods will be compared, using samples that were previously analyzed by NGS.

The goal of the study is to assess whether MS can represent or not a faster and cheaper way to detect key point mutations in patients suffering from hematological malignancies

ELIGIBILITY:
Inclusion Criteria:

* adults >18 years old
* anonymized samples already studied with NGS in Strasbourg university hematology center for somatic mutations
* non-opposition of the patient for testing the archive sample with the new method

Exclusion Criteria:

* opposition for testing the archive sample with the new method
* insufficient archival material
* patient under protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: anonymized samples from patients already studied with NGS in Strasbourg university hematology center for somatic mutations
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Detection of somatic mutations in hematological malignancies by using mass spectrometry (MS) | 10 months
  Detection of somatic mutations in hematological malignancies is now routinely assessed by NGS sequencing. This powerful approach is nevertheless time consuming and its costs represent limitation for its availability. An original approach is now available, using mass spectrometry (MS). In this study the analytical performance of both methods will be compared, using samples that were previously analyzed by NGS.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MAUVIEUX, MD, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Laboratoire d'Hématologie, Strasbourg, France